CLINICAL TRIAL: NCT06700044
Title: Assessing the Effects of Probiotic Supplementation in Women With High-Risk Pregnancies: A Randomized Controlled Trial
Brief Title: Probiotic Supplementation During Pregnancy in Women With High-Risk Pregnancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: ImmuneBiotech Medical Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dnr 2024-03036-02
Record Dates: First submitted 2024-10-10; First posted 2024-11-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Preeclampsia; Gut Dysbiosis
Keywords: preeclampsia; probiotics; microbiome; lactobacillus; pregnancy; GutMagnific
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-risk probiotic (Active Comparator): 50 pregnant women with high risk of developing PE will take one stick/10^9 CFU of probiotic dietary supplement GutMagnific per day from gestational week 12 until partus.
  Interventions: Dietary Supplement: GutMagnific
- High-risk placebo (Placebo Comparator): 50 pregnant women with high risk of developing PE will take one stick/placebo per day from gestational week 12 until partus.
  Interventions: Dietary Supplement: Placebo
- Low-risk probiotic (Active Comparator): 25 pregnant women with low risk of developing PE will take one stick/10^9 CFU of probiotic dietary supplement GutMagnific per day from gestational week 12 until partus.
  Interventions: Dietary Supplement: GutMagnific
- Low-risk placebo (Placebo Comparator): 25 pregnant women with low risk of developing PE will take one stick/placebo per day from gestational week 12 until partus.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GutMagnific — Participants will take one stick/10^9 CFU of probiotic dietary supplement GutMagnific per day from gestational week 12 until gestational week 37
  Arms: High-risk probiotic; Low-risk probiotic
Dietary Supplement: Placebo — Participants will take one stick/placebo per day from gestational week 12 until partus.
  Arms: High-risk placebo; Low-risk placebo

SUMMARY:
Preeclampsia (PE) is a complication during pregnancy characterized by hypertension, organ damage, and inflammation, without an effective treatment. The underlying mechanisms causing the disease also remain partly unknown. In this double-blind placebo-controlled study, the effects of probiotic dietary supplement GutMagnific during pregnancy will be assessed in pregnancies with a high risk of PE as well as low risk. The hypothesis is that probiotic dietary supplement GutMagnific can prevent or reduce the inflammatory response and clinical manifestations associated with PE through counteracting imbalances in the oral and gut microbiome composition.

DETAILED DESCRIPTION:
PE is a leading cause of maternal and fetal morbidity and mortality worldwide, affecting 3-7% of pregnant women. PE is characterized by hypertension and organ damage manifesting after 20 gestational weeks, and is associated with an increased systemic inflammatory response in the mother. The clinical manifestations may vary greatly and are often more severe in early-onset PE (onset <34 gestational weeks) than late-onset PE (onset ≥34 gestational weeks). Severe features include blood-pressure ≥160/110 mmHg, severe organ dysfunction, stroke, and eclampsia. Placental failure is central in the pathophysiology of PE, although the underlying mechanisms causing the disease remain partly unknown. Current research, including a previous study conducted by the investigators, suggests that disturbances in the gut microbiome might be involved in the pathogenesis of PE, leading to a dysfunctional immune response and damaged gut barrier functions. The investigators' previous study also indicated that PE is associated with gastrointestinal symptoms.

GutMagnific is an evidence-based probiotic dietary supplement, shown to be effective in correcting disturbances in the gut microbiome, reduce inflammation and repair a damaged gut barrier. It was originally developed for treatment of irritable bowel syndrome (IBS). There is an overlap in immunological responses involved in PE and IBS, and women with IBS have a higher risk of developing PE. Therefore, the investigators expect that the product might also have positive effects in pregnant women with a high risk of PE.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 18 years old
* High risk of PE (≥ 1 high-risk factor, or ≥3 moderate risk factors according to the Swedish Society of Obstetrics and Gynecology (SFOG) 2019 guidelines); or low risk of PE (no high-risk factors, or <3 moderate risk factors):

  * High risk factors are:

    * Auto-immune diseases such as SLE or anti-phospholipid syndrome
    * Previous preeclampsia or eclampsia
    * Previous hypertension of pregnancy with preterm birth before gestational week 34, growth restriction, intrauterine fetal death or ablatio
    * Type 1 or 2 diabetes
    * Duplex (or triplex) pregnancy
    * Kidney disease
    * Chronic hypertension
    * IVF with egg donation
  * Moderate risk factors are:

    * Nulliparity
    * Heredity for preeclampsia (at least one of mother, maternal grandmother, or sister)
    * BMI>30
    * Age>40
    * Pregnancy interval >10 years
    * Systolic blood pressure >130 mmHg or diastolic blood pressure > 80 mmHg at admission in antenatal maternity care
    * African descent
    * Verified obstructive sleep apnea
* Ability to give written informed consent

Exclusion Criteria:

* Enrollment in another clinical study
* Use of other probiotic supplements in the last 2 weeks before baseline, or during the course of the study
* Use of antibiotics in the last 6 weeks
* Current treatment with metformin, progesterone, or regular medical treatment which may impact study aim (e.g. laxatives)
* Immunosuppression
* Diabetes mellitus (type I and type II)
* Inflammatory bowel disease
* Celiac disease
* Bad obstetric history
* Other serious conditions that might affect gut flora or capability of the subject to participate
* Language difficulties or difficulties understanding informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in oral and gut microbiota composition | Around gestational week 12 (baseline), 28, 37, and 6-8 weeks postpartum. In the event of a participant developing PE, samples will be taken at PE diagnosis as well.
  Fecal and salivary samples will be analyzed using next-generation sequencing techniques to monitor possible changes related to probiotic supplement, and possible associations with obstetric outcome (especially PE incidence) will be assessed. Samples taken prior to, during and after probiotic treatment in the same participant will be compared.

SECONDARY OUTCOMES:
Changes in gastrointestinal symptoms | At the baseline and every two weeks until 6-8 weeks postpartum.
  A modified questionnaire for irritable bowel syndrome (IBS) symptoms will be filled in by participants grading different gastrointestinal symptoms from 1-10. Higher score indicates better condition.
Changes in blood pressure | At the baseline and continuously every 2-3 weeks from gestational week 24 throughout the pregnancy, and 6-8 weeks postpartum.
  Blood pressure measurements at standard midwife appointments in antenatal care.
Differences in obstetric outcome | Data will be collected from the Swedish Pregnancy Register (Graviditetsregistret) and/or medical records through study completion, an average of 6 months for term pregnancies.
  Incidence of adverse events during pregnancy, including PE, fetal growth restriction, gestational hypertension, gestational diabetes mellitus, and preterm birth.
Changes in oral glucose tolerance test results | Gestational week 28
  Blood glucose levels before (fasting) and after standard oral glucose tolerance test will be assessed to study possible effects of probiotic supplementation.
Changes in circulatory Short-chain fatty acids (SCFAs) levels | Around gestational week 12 (baseline), 28, 37, and 6-8 weeks postpartum. In the event of a participant developing PE, samples will be taken at PE diagnosis as well.
  Analysis of SCFAs levels in blood samples will be assessed to study possible effects of probiotic supplementation.
Changes in circulatory Lipopolysaccharide (LPS) levels | Around gestational week 12 (baseline), 28, 37, and 6-8 weeks postpartum. In the event of a participant developing PE, samples will be taken at PE diagnosis as well.
  Analysis of LPS levels in blood samples will be assessed to study possible effects of probiotic supplementation.
Changes in metabolic parameters | Around gestational week 12 (baseline), 28, 37, and 6-8 weeks postpartum. In the event of a participant developing PE, samples will be taken at PE diagnosis as well.
  Analysis of metabolic parameters such as ferritin will be assessed to study possible effects of probiotic supplementation.
Change in systemic cytokine levels | Around gestational week 12 (baseline), 28, 37, and 6-8 weeks postpartum. In the event of a participant developing PE, samples will be taken at PE diagnosis as well.
  Cytokines relevant in PE including IL6, IL1, IL10, IL17, TNF-alfa and interferon-gamma will be measured in blood samples to monitor possible effects of probiotic supplementation on the maternal inflammatory response.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skåne, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No